CLINICAL TRIAL: NCT05834985
Title: Endoscopic Management Of Controlled Colo-cutaneous Fistula As A Complication of Acute Sigmoid Diverticulitis: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mohamed Shehata
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Fistula; Sigmoid
Keywords: stent, endoscopy , enod-stitches, diverticulitis
MeSH Terms: conditions — Fistula; Diverticulitis

STUDY DESIGN:
Intervention Model Description: The investigators included all patients who were presented to General Surgery Department with Controlled Colo-cutaneous Fistula As A complication of Acute Diverticulitis at Zagazig University hospital between (December 2020 to April 2023). the calculated sample size equal 66 patients divided into two equal groups. Included patients were randomized at a 1:1 ratio to "Endoscopic Group, EG" or "Surgical Group , SG" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention.(simple random sample). Patients will be divided into 2 groups in accordance type of preoperative
  Therapy :
  Group 1: "Endoscopic Group, EG" included 33 patients. Group 2: "Surgical Group , SG" included 33 patients.
  Inclusion criteria:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) endoscopic group (Active Comparator): For patients in EG, we began with assessment of the site & size of fistula . In this study, OTSC was used in 9 patients .We started deploying the clips perpendicular to the long axis of the defect. If needed, more than one clip was sequentially deployed, starting at edge of the defect towards the center. Standard clips were passed through-the-scope to achieve superficial tissue apposition engaging the mucosa and submucosa (with 1.2-mm-wide and 6-mm-long arms capable of an approximately 12-mm grasp) and were used in conjunction with thermal ablation or mechanical scraping of the tissue around the edges of the defect to achieve a more resilient seal.
  Concurrently, the interventional radiology team subcutaneously drained the intraperitoneal free fluid using 2 intra-peritoneal tubes that were placed under US guidance in the sub-hepatic region and in the pelvis
  Interventions: Procedure: endoscopic management of fistula due to sigmoid diverticulitis by clip or endostitches
- group (2) surgical group (No Intervention): sigmoid resection after proper colonic preparation with primary anstomosis with circular stapler either open or laparoscopically

INTERVENTIONS:
Procedure: endoscopic management of fistula due to sigmoid diverticulitis by clip or endostitches — endoscopic management of fistula due to sigmoid diverticulitis by clip or endostitches
  Arms: group (1) endoscopic group

SUMMARY:
Diverticular disease is a common condition in western countries with relatively uncommon complications[1]. Fistulae complicating diverticulitis are the result of a localized perforation into adjacent viscera, and occur in 4-23% of patients hospitalized for diverticular disease[2]. The types of fistulae include colovesical, colovaginal, colotubal, coloenteric, and colocutaneous fistulae[3]. Colocutaneous fistulae occur very rarely, accounting for 1-4% of the total number of fistulae complicating colonic diverticular disease[4]. Herein we describe a case of a fistula connecting the sigmoid colon with the left flank-lower lumbar area, due to diverticulitis of the sigmoid colon[5].

A new over-the-scope clip system, called OTSC (Ovesco Endoscopy, Tübingen, Germany), appeared on the market about 3 years ago[6]. The system consists of a nitinol clip loaded at the tip of the endoscope that can capture a large amount of tissue and compress the lesion until healed[7]. Results from animal models and initial clinical use support the efficacy of OTSC closure in the treatment of gastrointestinal bleeding; its role in the management of iatrogenic perforations in humans is less defined, and reports on its use in treating colorectal postsurgical leaks and fistulas are anecdotal [8]. Here we report on the use of OTSC in the endoscopic treatment of colo-cutaneous fistula as acomplication of acute diverticultis .

DETAILED DESCRIPTION:
Diverticular disease is a common condition in western countries with relatively uncommon complications[1]. Fistulae complicating diverticulitis are the result of a localized perforation into adjacent viscera, and occur in 4-23% of patients hospitalized for diverticular disease[2]. The types of fistulae include colovesical, colovaginal, colotubal, coloenteric, and colocutaneous fistulae[3]. Colocutaneous fistulae occur very rarely, accounting for 1-4% of the total number of fistulae complicating colonic diverticular disease[4]. Herein we describe a case of a fistula connecting the sigmoid colon with the left flank-lower lumbar area, due to diverticulitis of the sigmoid colon[5].

A new over-the-scope clip system, called OTSC (Ovesco Endoscopy, Tübingen, Germany), appeared on the market about 3 years ago[6]. The system consists of a nitinol clip loaded at the tip of the endoscope that can capture a large amount of tissue and compress the lesion until healed[7]. Results from animal models and initial clinical use support the efficacy of OTSC closure in the treatment of gastrointestinal bleeding; its role in the management of iatrogenic perforations in humans is less defined, and reports on its use in treating colorectal postsurgical leaks and fistulas are anecdotal [8]. Here we report on the use of OTSC in the endoscopic treatment of colo-cutaneous fistula as acomplication of acute diverticultis .

Rationale:

As endoscopy is less invasive maneuver and can be done without general anathesia , so we will try to close the fistula due to acute diverticulitis with OVASCO clip , to avoid major surgery with also high incidence of recurrence again . there is only one clinical trial for this resons , so we will try to achieve result to concolude the use of endoscopy in management GIT fistulas.

Research question:

Is Endoscopic Management Of Controlled Colo-cutaneous Fistula As A complication of Acute Diverticulitis Effective?

Hypothesis:

Yes The Endoscopic Management Of Low Output Recurrent Colonic Fistula After Anterior Resection For Rectal Cancer Is Effective .

Aim of the work

Management Of Controlled Colo-cutaneous Fistula As A complication of Acute Diverticulitis & reducing the morbidity & mortality Endoscoplically.

Objectives

1. To evaluate the advantages and safety of Endoscopic Management Of Controlled Colo-cutaneous Fistula As A complication of Acute Diverticulitis.
2. To evaluate the effect of Endoscopic Management Of Controlled Colo-cutaneous Fistula As A complication of Acute Diverticulitis in reducing morbidity and postoperative hospital stay.

Subjects and Methods

Technical design:

A- Site of the study: The investigators included all patients who were presented to General Surgery Department with Controlled Colo-cutaneous Fistula As A complication of Acute Diverticulitis at Zagazig University hospital between (December 2020 to August 2023).

B- Sample size:

The sample size was calculated by using open Epi program depending on the following data ; confidence interval 95% , power of the test 80% , ratio of unexposed/ exposed 1 , the success rate of surgical repair versus endoscopic repair was 89 % versus 71 % respectively. Odd ratio 3.3 , and risk ratio 1.3 , so the calculated sample size equal 66 patients divided into two equal groups.

c- Sample selection: Included patients were randomized at a 1:1 ratio to "Endoscopic Group, EG" or "Surgical Group , SG" via the drawing of sealed envelopes containing computer-generated random numbers prepared by a third party before the start of the intervention.(simple random sample).

D- Subjects: Patients will be divided into 2 groups in accordance type of preoperative

Therapy :

Group 1: "Endoscopic Group, EG" included 33 patients. Group 2: "Surgical Group , SG" included 33 patients.

Inclusion criteria:

Patients with Controlled Colo-cutaneous Fistula As A complication of Acute Diverticulitis , recurrent fistula , failued conservative meaures .patient with good general condition (ASA I&II).

Exclusion criteria:

We excluded patients who bad general condition (ASAIII&IV&V), patients with high output fistula , respond to conservative measures.

E- Data collection (tools): All patients will subjected to the followings:

patients were selected by randomization method, full history taking, Complete physical examination, laboratory investigations (complete blood picture, liver and kidney functions, coagulation profile, tumor marker tests, serum electrolytes), patients were assessed radio-logically by abdominal x- ray , abdominal ultrasound, pelvic and abdominal CT.

Study design (operational study):

A. Type of the study : A randomized Controlled Trial.

B. Steps of performance:

1. Complete history taking.
2. Clinical and laboratory results.
3. Radiological results.
4. Endoscopic management of Controlled Colo-cutaneous Fistula As A complication of Acute Diverticulitis.
5. Analysis of the results.
6. Preparing conclusion and recommendation.

C-Study techniques (procedure):

For patients in EG, we began with assessment of the site & size of fistula . In this study, OTSC was used in 9 patients .We started deploying the clips perpendicular to the long axis of the defect. If needed, more than one clip was sequentially deployed, starting at edge of the defect towards the center. Standard clips were passed through-the-scope to achieve superficial tissue apposition engaging the mucosa and submucosa (with 1.2-mm-wide and 6-mm-long arms capable of an approximately 12-mm grasp) and were used in conjunction with thermal ablation or mechanical scraping of the tissue around the edges of the defect to achieve a more resilient seal.

Concurrently, the interventional radiology team subcutaneously drained the intraperitoneal free fluid using 2 intra-peritoneal tubes that were placed under US guidance in the sub-hepatic region and in the pelvis.

D-Outcomes:

Primary and secondary outcomes were incidence of postoperative hospital stay and complications in each group during the 3-months follow-up period, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Controlled Colo-cutaneous Fistula As A complication of Acute Diverticulitis , recurrent fistula.
* failued conservative meaures .
* patient with good general condition (ASA I&II).

Exclusion Criteria:

* We excluded patients who bad general condition (ASAIII&IV&V),
* patients with high output fistula ,
* respond to conservative measures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
incidence of recurrence of fistula | within one week after the endoscopy
  incidence of recurrence of fistula

SECONDARY OUTCOMES:
incidence of side effects of endoscopy | within one month after the surgery
  incidence of side effects of endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, MD, Principal Investigator — ZAGAZIG UNIVERSITY HOSPITALS
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqua, Egypt

IPD SHARING:
Plan to Share IPD: No